CLINICAL TRIAL: NCT01872546
Title: Skin Transcriptional Profiles In Psoriatic Patients Under Adalimumab Biotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CYTOPSO
Record Dates: First submitted 2013-03-27; First posted 2013-06-07 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Plaque Psoriasis
MeSH Terms: interventions — Adalimumab

ARMS (1):
- Adalimumab (Experimental)
  Interventions: Drug: HUMIRA 40mg

INTERVENTIONS:
Drug: HUMIRA 40mg

SUMMARY:
The expertise in the characterization of transcriptomics profile in lesional psoriatic skin and on the availability of innovative therapy for these patients.The investigators propose to follow the modification of the skin transcriptomics profile in psoriatic patients during successful Adalimumab biotherapy. Skin transcriptomics profiles of normal skin, psoriatic non lesional skin, and psoriatic lesional skin before and after biotherapy will be compared. The investigators will focus on the modification of the cytokine "signature" in these skin lesions and of some markers of keratinocyte inflammation. The modification of the transcriptomics profile induced by the biotherapy will be correlated to the clinical response Psoriasis Area and Severity Index.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic plaque psoriasis involving at least 10% of body surface area with no previous biotherapy.
* Adalimumab prescribed in usual practice

Exclusion Criteria:

* Patients presenting a contraindication to the use of Adalimumab:

hypersensibility in Adalimumab or in one of the excipients.

* Patients presenting an evolutionary tuberculosis or the other severe infections such as sepsis and opportunist infections
* presenting patients one cardiac insufficiencies moderated in severe
* Patients under anakinra or abatacept
* current participation in another study of clinical research

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Analyze modifications of the skin inflammatory | 1 month
  comparaison skin biopsy in non-lesional area between skin biopsy lesional area

SECONDARY OUTCOMES:
skin transcriptomic profile | 1 month
  5 mL blood sample for serum preparation

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Poitiers, Poitiers, France